CLINICAL TRIAL: NCT02905708
Title: Efficacy Warming Garment to Maintain Normothermia Using Integrated Chemical Heat Pack Construction, in the Perioperative Period, for Surgery Less Than 12 Hours Duration
Brief Title: Efficacy of Warming Garment in the Perioperative Period With Integrated Chemical Heat Packs to Maintain Normothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr K Services PC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DrKirwan IRB#16-11
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Hypothermia
Keywords: normothermia; hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Forced Air Warming Device (Active Comparator): Active Comparator: Forced Air Warming Device first group will have the warming devices started in the pre-operative area. You will receive a full body forced air warming. Device is non experimental and FDA approved, used within the hospital to keep patients warm.You will then have your temperature taken and documented by the staff at various prescribed times.
  Warming in the operating room: You will receive the same or a similar warming device known as a Bair Hugger and warmed IV fluids once you are in the operating room. Bair Paws or Bair Hugger will also be used in the post-anesthesia care area.
  Interventions: Device: Forced Air Warming Device
- Air-Activated heating packs (Active Comparator): The second group will receive the study warming device which consists of a jacket, pants, gloves and socks with integrated Air-Activated heating packs. Device is supplied vacuum packed, heat packs of iron powder/activated charcoal activated by air. Device applied at least twenty minutes prior to surgery. The same device will be maintained in place throughout the surgery and the post-anesthesia period.
  Interventions: Device: Air-Activated heating packs

INTERVENTIONS:
Device: Air-Activated heating packs — The subject disrobe and will dress in a jacket, pants, gloves and socks (ensemble) which will be removed from a vacuum pack. He will be assisted by the nurse in pre-operative area. The ensemble will remain in place until the subject is fully recovered from anesthesia.
  Other Names: Garment with heat packs - iron powder and activated charcoal
  Arms: Air-Activated heating packs
Device: Forced Air Warming Device — forced air-warming inflatable device applied according to standard hospital protocol.
  Other Names: forced air-warming device
  Arms: Forced Air Warming Device

SUMMARY:
Efficacy of Stand-alone, Non-tethered, Self-applying Warming Garment in the Preoperative, Intraoperative and Postoperative Recovery Period; Using an Integrated Chemical Heat Pack Construction, With a View to Maintaining Normothermia During the Peri-operative Period

DETAILED DESCRIPTION:
Subjects will be randomized into two groups. The first group will have the standard warming devices currently used which consists of a forced air warming device. This will be applied in the form of a gown in the pre-operative area. The device is called the Bair Paws. (Subjects will either continue with this or have a separate forced air warming device applied in the operating room called a Bair Hugger.) This device is non experimental and is FDA approved and used within the hospital to keep patients warm. They will then have their temperature taken and documented by the staff at various prescribed times.

The second group will receive the warming devices being studied which consist of a jacket, pants, gloves and socks with integrated air-activated chemical heat packs. The garment is applied at least twenty minutes prior to surgery. The same warming device will be maintained in place throughout the surgery and the period of post-anesthesia.

Intraoperative period: The participants temperature will be monitored and documented at prescribed times.

Postoperative period: The participants will have temperature monitored in the post anesthesia care area. Your part in this study will last until you are admitted to your room after surgery or you change into your own clothes prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

Male Female ASA physical status classification system Class I ASA physical status classification system Class II Age 18-80

Exclusion Criteria:

ASA physical status classification system Class III -VI Body Mass Index greater than 37.0

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Core body temperature, degrees Centigrade | Peri-operative period - 15 minutes before surgery to 4 hours after termination of surgery.
  Measurement of core body temperature, degrees Centigrade, 15 minutes intervals during above time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence A Kirwan, M.D., Principal Investigator — Dr. K. Services P.C.
Locations (1):
- Norwalk Hospital, Norwalk, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brandt S, Oguz R, Huttner H, Waglechner G, Chiari A, Greif R, Kurz A, Kimberger O. Resistive-polymer versus forced-air warming: comparable efficacy in orthopedic patients. Anesth Analg. 2010 Mar 1;110(3):834-8. doi: 10.1213/ANE.0b013e3181cb3f5f. Epub 2009 Dec 30. PMID 20042442